CLINICAL TRIAL: NCT03558009
Title: Epidemiological Analysis for Hereditary Angioedema Disease: An International, Multicenter, Epidemiological Protocol
Brief Title: Epidemiological Analysis for Hereditary Angioedema Disease
Acronym: EHA
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: EHA 01-2018
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Abdominal Pain; Functional Abdominal Pain
Keywords: Hereditary Angioedema; DBS-based biochemical and genetic assay for HAE type I/II; Biomarker
MeSH Terms: conditions — Abdominal Pain; Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with abdominal pain attacks: Participants experiencing recurrent abdominal pain attacks without a clear etiolgy aged between 2-60 years

SUMMARY:
An international, multicenter, epidemiological, observational study investigating the prevalence of Hereditary Angioedema (HAE) disease among participants with recurrent episodes of abdominal pain of no obvious etiology.

DETAILED DESCRIPTION:
Hereditary Angioedema (HAE) is a rare autosomal dominant disorder characterized most commonly by deficient (type 1) or nonfunctional (type 2) C1 inhibitor protein (encoded by SERPING1 gene). The disorder is associated with episodes of angioedema of the face, larynx, lips, abdomen, and extremities. The angioedema is caused by the activation of the kallikrein-kinin system that leads to the release of vasoactive peptides, followed by edema, which in severe cases can be life threatening.

Gastrointestinal involvement occurs in 93% of patients with HAE and may be the only manifestation of the disease. However, individuals with gastrointestinal symptoms are rarely considered for HAE and the disease can be misdiagnosed for several years.

EHA study focuses on the gastrointestinal complications of HAE as a potential area of misdiagnosis leading to surgical morbidity. Aim of the study is to investigate the prevalence of HAE among participants experiencing recurrent abdominal pain attacks with no clear etiology. The HAE-positive samples in the study will be further analyzed biochemically to identify disease-specific biomarker that may support the development of new diagnostic tools for HAE disease.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent will be obtained from the participant or the parent or legal guardian
* Participants with previous episodes of abdominal pain of no obvious etiology
* Participants aged between 2 to 60 years old

EXCLUSION CRITERIA

* Previous diagnosis of HAE
* Inability to provide informed consent
* The etiology of abdominal pain attacks is determined
* Participants that are younger than 2 years old or older than 60 years old
* Previous enrolled in the study

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with previous episodes of abdominal pain attacks of no obvious etiology
Sampling Method: Probability Sample
Enrollment: 2318 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Epidemiological analysis of prevalence of the HAE in participants with previous episodes of abdominal pain of no obvious etiology. | 4 years
  Dry Blood Spot (DBS)-based biochemical measurements of C4 complement and the protease C1 inhibitor levels will be analyzed via liquid chromatography multiple reaction. The pathological biochemical results will be genetically validated via combination of the Next-Generation Sequencing (the mutation will be confirmed by Sanger sequencing) and Multiplex ligation-dependent probe amplification of SERPING1.

SECONDARY OUTCOMES:
Establishment of a biomarker in HAE-positive cohort | 4 years
  HAE-positive samples will be analyzed for the identification of potential biomarkers (based on MS/MS-Tandem spectroscopy) and compared with the merged control samples in order establish a HAE specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, MD, Study Chair — CENTOGENE GmbH
Locations (35):
- Germany (8):
  - Praxis und Tagesklinik Prof. Dr. med. Jens Papke, Neustadt, Saxony
  - Universitätsklinikum Düsseldorf, Klinik für Allgemein-, Viszeral- und Kinderchirurgie, Düsseldorf
  - Dr. med. Engelhard | Dr. med. Wihl, Internistische Gemeinschaftspraxis, Frankenberg
  - Universitätsmedizin Greifswald Körperschaft des öffentlichen Rechts, Greifswald
  - Klinikum Kassel GmbH, Kassel
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Johannes Wesling Klinikum Minden, Universitätsklinik der Ruhr Universität Bochum, Minden
  - Kinder- und Jugendklinik, Universitätsmedizin Rostock, Rostock
- Azienda Ospedaliera Antonio Cardarelli, Napoli, Italy
- Hiroshima University Graduate School of Biomedical Sciences, Hiroshima, Japan
- Poland (8):
  - Gastromed, Bialystok
  - Centrum Medyczne Alfamedica Silesia North, Częstochowa
  - Specialized Medical Offices MeaMedica, Gdansk
  - Przychodnia Polskiej Fundacji Gastroenterologii, Warsaw
  - WIP Warsaw IBD Point, Warsaw
  - Przychodnia Lekarska MediSpace, Warsaw
  - Uniwersytecki Szpital Kliniczny, Wroclaw
  - Cdl "Barska", Włocławek
- Turkey (Türkiye) (4):
  - Cukurova University Balcali Hospital, Adana
  - Bezmialem Vakif Üniversitesi, Istanbul
  - Ege University Faculty of Medicine, Izmir
  - Dokuz Eylül University Research and Application Hospital, Izmir
- United Kingdom (13):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospital of Derby and Burton NHS Foundation Trust, Derby
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Alexandra Hospital, Glasgow
  - University Hospital Crosshouse, Kilmarnock
  - University Hospital Leicester (UHL), Leicester
  - The Royal London Hospital, London
  - St Thomas Hospital, London
  - St George's University Hospital London, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester Royal Infirmary, Manchester
  - Milton Keynes Hospital, Milton Keynes